CLINICAL TRIAL: NCT01211899
Title: Incidence and Prognosis of Disseminated Intravscular Coagulation in Patients Severe Sepsis and Septic Shock; Association With 4G/5G Polymorphism of PAI-1 Gene
Brief Title: 4G/5G Polymorphism of Plasminogen Activator Inhibitor-1 Gene and Disseminated Intravascular Coagulation in Severe Sepsis and Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: f2000tj2
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Severe Sepsis
Keywords: polymorphism,; plasminogen activator inhibitor,; disseminated intravascular coagulation,
MeSH Terms: conditions — Sepsis; Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for 4G/5G polymorphism of plasminogen activator inhibitor-1 (PAI-1)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Data on 4G/5G polymorphism of plasminogen activator inhibitor-1 (PAI-1) gene are limited in Asian patients with sepsis. Therefore, the investigators aim to prospectively investigate the incidence of 4G/5G polymorphism and its relationship with disseminated intravascluar coagulatin in patients with severe sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult patinents aged > 18 years, Patients satisfying the criteria by 2008 Surviving Sepsis Campagin, Patients who are determined as having a sepsis within 24 hours of ICU stay

Exclusion Criteria:

* Do-not-resuscitate, cardiopulmonary resuscitation, ICU stay < 1 day, Refusal to participate in the study, Hematologic malignancy or liver cirrhosis (Child C), Congenital abnormality in coagulation system, Transfer from other ICUs or hospitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU for severe sepsis or septic shock
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated)